CLINICAL TRIAL: NCT01251666
Title: Comparison of Performances of Two Automated Immunochemical Faecal Occult Blood Tests in Colorectal Cancer Screening, in Reference to Usual Care Guaiac Test
Brief Title: Comparison of Hemoccult, Magstream and OC-Sensor Faecal Occult Blood Tests in Colorectal Cancer Screening
Acronym: HeMO
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Caen (Other)
Collaborators: National Cancer Institute, France (Other Government); Ligue contre le cancer, France (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Double | Purpose: Screening
Other Study IDs: 2008-A01463-52
Record Dates: First submitted 2010-11-29; First posted 2010-12-02 (Estimated); Last update posted 2012-09-03 (Estimated); Status verified 2012-08

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Screening; Average-risk population; faecal occult blood tests
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Colonoscopy

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Magstream + Oc Sensor + Hemoccult II (Other): Each patient will perform all three tests:
  * Magstream: 2 samples (each on a different stool)
  * OC Sensor: 2 samples (each on a different stool)
  * Hemoccult II: 6 samples (2 samples per stool, on 3 different stools)
  Each test will be considered as positive if at least one sample is positive (cutoff for Magstream 55 ng/ml and for OC Sensor 150 ng/ml).
  Screening will be considered as positive if at least one of the three tests is positive, leading to a colonoscopy
  Interventions: Other: Colonoscopy

INTERVENTIONS:
Other: Colonoscopy — Colonoscopy if at least one of the faecal occult blood tests is positive (blinded to each test result)

SUMMARY:
Colorectal cancer screening by faecal occult blood test (FOBT) is a high public health priority. The interest of guaiac tests (G-FOBT) is limited by their poor sensitivity, while the superiority of I-FOBT in comparison with G-FOBT is now established. Nevertheless automated quantitative I-FOBTs have not been compared, and the optimal number of samples and threshold is not yet fixed. The aim of this study is to compare the performances of the 2 more well-known I-FOBTs with automated analyzers (magstream by Fujirebio, and OC Sensor by Eiken) for different positivity thresholds and numbers of samples in general average risk population. Patients will performed a two samples Magstream, a two samples OC Sensor and Hemoccult II. In case of a positive test, a colonoscopy will be performed. Sensitivity and specificity for detection of cancer and advanced neoplasias will be compared between tests using ratio of sensitivities (RSN) and ratio of false positives (RFP) according to number of samples and positivity threshold.

ELIGIBILITY:
Inclusion Criteria:

* 50 to 74 years
* Informed consent signed

Exclusion Criteria:

* Recent digestive symptoms
* Complete colonoscopy less than 5 years ago
* Personal history of colorectal cancer or colorectal adenoma or colonic disease requiring regular colonoscopy surveillance
* Familial history of colorectal cancer in a first degree next of kin before 65 years, or two cases in first degree next of kin.
* Severe extra-intestinal disease
* Screening ill-timed (ex. depression)

Ages: 50 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 19797 (Actual)
Dates: Start 2008-06; Primary Completion 2012-06 (Actual); Study Completion 2012-08 (Actual)

PRIMARY OUTCOMES:
Ratio of sensitivities (RSN) for detection of advanced neoplasias | Up to 6 months after faecal occult blood test (FOBT) (At the time of colonoscopy)
  Advanced neoplasias included invasive cancers and high-risk adenomas (larger than 1 cm or with high grade dysplasia).
  RSN is the ratio of the true positives of two tests. True positives for one test are patients positive for the test, with targeted lesion (here advanced neoplasias).
  RSN will be calculed between immunochemical tests, and for each immunochemical test in reference to gaiac test.

SECONDARY OUTCOMES:
Ratio of False Positives (RFP) for detection of invasive cancers | Up to 6 months after FOBT (At the time of colonoscopy)
  RFP is related to specificity. False positives of one test are patients with a positive test but without targeted lesions (here invasive cancers).
  RFP will be calculed between immunochemical tests, and for each immunochemical test in reference to gaiac test.
RFP for detection of advanced neoplasias | Up to 6 months after FOBT (At the time of colonoscopy)
  RFP is related to specificity. False positives of one test are patients with a positive test but without targeted lesions (here advanced neoplasias).
  RFP will be calculed between immunochemical tests, and for each immunochemical test in reference to gaiac test.
Relative Receiver Operating Characteristics(ROC) curves | Up to 6 months after FOBT (At the time of colonoscopy)
  Relative ROC curves plots RSN according to RFP (similar to ROC curve). Relative ROC curves will be compared in reference to gaiac test, according to number of samples analysed for each immunochemical test, and the way they are analysed.
Detection rate of invasive cancer | Up to 6 months after FOBT (At the time of colonoscopy)
Detection rate of advanced neoplasias | Up to 6 months after FOBT (At the time of colonoscopy)
Cost-effectiveness analysis | Up to 6 months after FOBT (At the time of colonoscopy)
  It will take into account number of samples and threshold
Predictive positive value for detection of invasive cancers | Up to 6 months after FOBT (At the time of colonoscopy)
Predictive value for detection of advanced neoplasias | Up to 6 months after FOBT (At the time of colonoscopy)
Positivity rate | Immediate (At the time of FOBT)

CONTACTS AND LOCATIONS:
Overall Officials: Guy LAUNOY, MD-PhD, Study Director — University Hospital, Caen
Locations (2):
- France (2):
  - ADECA, Moulins
  - Adoc18 - Irsa, Saint-Doulchard

REFERENCES:
- [Derived] Raginel T, Puvinel J, Ferrand O, Bouvier V, Levillain R, Ruiz A, Lantieri O, Launoy G, Guittet L. A population-based comparison of immunochemical fecal occult blood tests for colorectal cancer screening. Gastroenterology. 2013 May;144(5):918-25. doi: 10.1053/j.gastro.2013.01.042. Epub 2013 Feb 1. PMID 23376426